CLINICAL TRIAL: NCT01009424
Title: A Multi-center, Placebo-controlled, Double Blind Multiple-ascending Dose Study in a Leapfrog Design to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of RO5024118 Following Repeated Inhalation in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease
Brief Title: A Multi-center Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of R7103 Following Repeated Inhalation in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NP22131
Record Dates: First submitted 2009-11-03; First posted 2009-11-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (6):
- 1 (Experimental): R7103 (dose 1) followed by placebo or placebo followed by R7103 (dose 1)
  Interventions: Drug: R7103
- 2 (Experimental): R7103 (dose 2) followed by placebo or placebo followed by R7103 (dose 2)
  Interventions: Drug: R7103
- 3 (Experimental): R7103 (dose 3) followed by placebo or placebo followed by R7103 (dose 3)
  Interventions: Drug: R7103
- 4 (Experimental): R7103 (dose 4) followed by placebo or placebo followed by R7103 (dose 4)
  Interventions: Drug: R7103
- 5 (Experimental): R7103 (dose 5) followed by placebo or placebo followed by R7103 (dose 5)
  Interventions: Drug: R7103
- 6 (Experimental): R7103 (dose 6) followed by placebo or placebo followed by R7103 (dose 6)
  Interventions: Drug: R7103

INTERVENTIONS:
Drug: R7103 — escalating inhaled dose

SUMMARY:
This study will assess the safety, tolerability, pharmacodynamics, and pharmacokinetics of RO5024118 following repeated inhalation in patients with moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD). Patients will be randomized to receive multiple inhaled doses of R7103, as compared with placebo. The target sample size is approximately 30 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 40-70 years of age, inclusive.
* Body Mass Index 18-32 kg/m2, inclusive.
* Female patients must be surgically sterile or post menopausal for the past year confirmed by a negative hormone panel. Male patients and their partners of childbearing potential must use two methods of contraception, one of which must be a barrier method for the duration of the study and for 7 days after last dose.
* Diagnosis of moderate-to-severe COPD (GOLD Stage II-III).

Exclusion Criteria:

* Current smoker or history of smoking in the last three months.
* Use of continuous daily long term oxygen therapy or requirement for oxygen therapy during exercise.
* History of cardiac conduction abnormalities or ventricular tachyarrhythmias.
* Exacerbation of COPD within 8 weeks before first dosing.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of multiple inhaled doses of R7103 as compared to placebo, and to define the Maximum Tolerated Dose (MTD) in target population | 18 days per arm

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche